CLINICAL TRIAL: NCT05776888
Title: Early Versus Late Ofatumumab (Kesimpta®) Use in Austrian RMS-Patients Over 2 Years- A Non-interventional Observational Study
Brief Title: Early Versus Late Ofatumumab (Kesimpta®) Use in Austrian RMS-Patients Over 2 Years
Acronym: KRONOS
Status: Active, not recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: COMB157GAT02
Record Dates: First submitted 2023-02-27; First posted 2023-03-20 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Relapsing Multiple Sclerosis
Keywords: relapsing multiple sclerosis; RMS; Ofatumumab; NIS
MeSH Terms: interventions — ofatumumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Early Treatment Cohort (Cohort 1): Patients that, before initiation of Ofatumumab, were either treatment naive or have started their treatment for RMS with another disease modifying therapy (BRACE, teriflunomide or fumarates). Non-naive patients in this cohort must have started the use of Ofatumumab within 3 years after first DMT initiation.
  Interventions: Other: Ofatumumab
- Later Treatment Cohort (Cohort 2): Patients that have been on BRACE and/or Teriflunomide and/or fumarates for at least three years or longer before the switch to Ofatumumab has been initiated.
  Interventions: Other: Ofatumumab

INTERVENTIONS:
Other: Ofatumumab — There is no treatment allocation. For both cohorts, only patients that have received Ofatumumab treatment for at least 3 months prior to inclusion in the study will be enrolled.

SUMMARY:
This non-interventional study aims to observe the effect of early versus late Ofatumumab treatment in RMS patients in a real-world setting in Austria over an observational period of 24 months.

DETAILED DESCRIPTION:
This multi-center, observational study will describe the effects of Ofatumumab in 2 cohorts in a routine medical care setting. Cohort one will comprise patients who have started Ofatumumab early during their disease (treatment naive patients or those that started Ofatumumab within 3 years of first therapy initiation). Cohort two will include patients who have been on other DMTs (one or several) for a minimum of 3 years prior to switching to Ofatumumab. Patients in both cohorts will be observed for two years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with relapsing multiple sclerosis (RMS) with disease activity defined by clinical assessment or MRI analysis.
2. Written informed consent must be obtained before participating in the study.
3. Patient is willing and able to complete the assessments, as outlined in this study.
4. Diagnosis of RMS per McDonald Criteria (2017) occurred prior to initiation of Ofatumumab.
5. Patients in both cohorts must have been on treatment with Ofatumumab for at least 3 months, but not longer than 12 months prior to inclusion in the study.
6. Cohort 1: Patients that, before initiation of Ofatumumab, were either treatment naive or have started their treatment for RMS with another disease modifying therapy (BRACE, teriflunomide or fumarates). Non-naive patients in this cohort must have started the use of Ofatumumab within 3 years after first DMT initiation.
7. Cohort 2: Patients must have been on either BRACE or Teriflunomide or fumarates for at least three years or longer before the switch to Ofatumumab has been initiated. Thus, this cohort includes patients that use Ofatumumab as second or later line DMT.

Exclusion Criteria:

1. Patients who have been on Ofatumumab less than 3 months or more than 12 months before inclusion.
2. Use of investigational drugs during the study, OR between Ofatumumab initiation and inclusion into the study, OR within 5 half-lives of investigational drug before Ofatumumab initiation, OR until the expected pharmacodynamic effect has returned to baseline, whichever is longer.
3. Use of any high efficacy therapy (including Fingolimod, Siponimod, Ponesimod, Ozanimod, Rituximab, Ocrelizumab, Natalizumab, Alemtuzumab, Mitoxantron or Cladribine) in either cohort prior to the initiation of Ofatumumab.
4. Previous use of any DMTs other than BRACE, Teriflunomide or fumarates prior to the initiation of Ofatumumab.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include male and female patients (aged ≥ 18 years) with a documented diagnosis of RMS and treated for at least 3 months with Ofatumumab
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients demonstrating NEDA-3 | from month 12 up to month 24
  Proportion and comparison of patients in both cohorts achieving NEDA-3 in the second year after treatment initiation, which refers to a comparison between month 12 and 24 after Ofatumumab treatment was initiated. NEDA-3 is defined by no confirmed MS relapse, no new or enlarging T2 lesions, no new Gadolinium-positive T1 lesions (in case Gadolinium was utilized), and no six-month confirmed disability worsening.

SECONDARY OUTCOMES:
Proportion of patients displaying NEDA-3, as well as individual NEDA components | Baseline, month 12, month 24
  Proportion of patients displaying NEDA-3, as well as individual NEDA components (i) experiencing no confirmed clinical relapses, (ii) lack of diseases progression measured by expanded disability status scale (EDSS) and (iii) absence of new disease activity (new or enhancing T2 or Gadolinium-positive T1 lesions (in case Gadolinium was utilized)), respectively, in the first treatment year (Baseline to month 12), the second treatment year (month 12 to month 24) as well as over the whole study period (Baseline to month 24).
Proportion of patients permanently discontinuing Ofatumumab during the study | Up to 24 months
  Proportion of patients permanently discontinuing Ofatumumab during the study, and reasons for discontinuation will be provided

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: No